CLINICAL TRIAL: NCT01527162
Title: Relationship of Orthotics to Activity and Participation in Children With Cerebral Palsy
Brief Title: Orthotics in Ambulatory Cerebral Palsy
Acronym: SAFO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Kristie Bjornson, Principal Investigator, Seattle Children's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: K23HD060764-03B; K23HD060764-03 (NIH)
Record Dates: First submitted 2012-01-30; First posted 2012-02-06 (Estimated); Results first posted 2016-02-04 (Estimated); Last update posted 2021-06-16 (Actual); Status verified 2021-05

CONDITIONS: Cerebral Palsy
Keywords: Cerebral palsy; orthotics; solid ankle foot orthoses
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SAFO worn (Experimental): Child wears their prescribed SAFO for 14 days
  Interventions: Device: SAFO worn; Other: SAFO not worn
- SAFO not worn (No Intervention): Child does not wear the prescribed SAFO for 14 days

INTERVENTIONS:
Device: SAFO worn — Child wears their prescribed SAFO for 14 days by random assignment
  Other Names: Solid ankle foot orthoses (SAFO)
  Arms: SAFO worn
Other: SAFO not worn — Child does not wear their prescirbed SAFO for 14 days by random assignment
  Other Names: Solid ankle foot orthoses (SAFO)
  Arms: SAFO worn

SUMMARY:
This project will examine the effect of solid ankle foot orthoses (SAFO) on day to day walking activity and life participation of ambulatory children with cerebral palsy. The investigators propose that SAFO have not effect on levels of walking and life participation versus not wearing the SAFO.

DETAILED DESCRIPTION:
This is a repeated measures trial with randomization of intervention in a cross over design which will quantify daily walking and physical activity levels for children with cerebral palsy (CP) with and without use of a solid ankle foot orthotic (SAFO). Current orthotic management guidelines are based primarily on evidence that SAFO use positively impacts body function and structure in clinic and lab based observations of activity and movement. Prior research has determined that wearing a SAFO improves different aspects of gait and mobility (stride and step length, single limb stance, velocity) for children with CP. However, these studies have been limited by small sample sizes, lack of comparison groups, inconsistency of orthotic fabrication, lack of clear and simple outcome measures and/or randomized control designs. No prior studies have evaluated the effect of SAFO use on activity performance outcomes.

The purpose of this study is to determine the effect of wearing or not wearing current SAFO on a child's walking ability, participation in common life activities, and gait. Children ages 2 - < 10 years who have bilateral cerebral palsy, dynamic equinus gait deformity, and wear bilateral SAFOs fabricated by Cascade DAFO will be approached for participation. Enrolled children are randomly assigned to either wear or not wear their SAFOs for a 14 day intervention period. After this period is over, children will then do the opposite for a second 14 day intervention period. Children attend three study visits; at enrollment, after the first intervention period is over, and after the second intervention period. At the first visit, parents and children (where applicable) complete questionnaires regarding their participation in common life activities in the prior 7 days, and complete a walking evaluation. Children wear a StepWatch accelerometer during each intervention period, which counts the number of steps the child takes and the time each step was taken. After the second intervention period is complete, the child's participation in the research study is complete. One home visit is conducted at the end of each intervention period, where the questionnaires are repeated, and the StepWatch is downloaded and/or re - calibrated per protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Age 2 to <10 years
2. Gross Motor Function Classification Scale Score of 1 - 3 (ambulatory)
3. Diagnosed with bilateral cerebral palsy
4. Has dynamic equinus gait deformity, defined as PROM to neutral, with equinus weight bearing pattern.
5. Wears bilateral SAFO more than 8 hours per day for more than one month.
6. Has a SAFO prescription of ankle at neutral (zero plantarflexion, with <10 degrees dorsiflexion).
7. The primary goal of the SAFO is to facilitate balance and walking
8. Has SAFOs fabricated by Cascade DAFO, Ferndale, WA.
9. Parent and child are willing to discontinue SAFO use for two weeks.

Exclusion Criteria:

1. Has visual impairment which limits physical activity.
2. Has had lower extremity Botox injections in the past 3 months.
3. Is expected to require changes to medications treating the movement disorder during the study period.
4. Has an uncontrolled seizure disorder which impacts mobility skills.
5. Has had neurosurgical or orthopedic surgeries in the past 6 months.
6. Has had other surgeries or procedures in the past two weeks.

Ages: 2 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2012-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristie Bjornson, PT, PhD, PCS, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Seattle Childrens Research Institute, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- SAFO Worn First, Then Not Worn: Child wears their prescribed SAFO for 14 days by random assignment and then not worn
- SAFO NOT Worn First, Then Worn: Child does not wear their prescirbed SAFO for 14 days by random assignment, then worn
Period: Overall Study
Arm/Group | SAFO Worn First, Then Not Worn | SAFO NOT Worn First, Then Worn
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: ages 3.0 to 5.8 years, mean age 4.3 years, spastic diplegia cerebral palsy, all wearing current AFO bilaterally to enhance walking activity
Groups:
- All Participants: We used a randomized cross-over design with eleven children with bilateral 9 CP, mean age 4.3 years. Subjects were randomized to their current SAFO worn or SAFO not worn for 2 weeks and then crossed over.
Arm/Group | All Participants
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 4.3 [3.0 to 5.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Walking Activity Levels
Description: Daily walking activity will be measured with the StepWatch accelerometer documenting average strides/day.
Time Frame: average of 5 days of second week of intervention
Measure: Mean (Standard Deviation); unit: average total strides/day
Arm/Group | SAFO Worn | SAFO Not Worn
Number analyzed (Participants) | 11 | 11
average total strides/day | 4660 (1421) | 4897 (1438)
Statistical Analysis 1: Comparison: SAFO Worn vs SAFO Not Worn; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Physical Activity Scale for Kids - Performance Version (ASKp)
Description: Physical activity will be by parental report of Physical Activities Scale for Kids performance version (ASKp) survey- total score. Scale ranges from 0 to 100 with higher scores representing more physical activity. A score of 100 on this criterion referenced evalutive measure is consistent with physical activity like that of a typically developing 5 year old.
Time Frame: previous 7 day reference
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SAFO Worn | SAFO Not Worn
Number analyzed (Participants) | 11 | 11
units on a scale | 51.08 (11.64) | 49.45 (14.2)
Statistical Analysis 1: Comparison: SAFO Worn vs SAFO Not Worn; Test type: Superiority or Other; p = 0.14, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Assessment of Life Habits for Children (LIFE-H)
Description: Participation in habits of daily life will be by parental report of the Life Habits questionnaire(Life-H for children) by the weighted total score on a scale of 0 to 9, with a higher score representing more participation in habits of daily life.
Time Frame: previous 7 day reference
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- SAFO Not Worn: Child does not wears their prescribed SAFO for 14 days
Arm/Group | SAFO Worn | SAFO Not Worn
Number analyzed (Participants) | 11 | 11
units on a scale | 5.71 (2.0) | 5.11 (2.2)
Statistical Analysis 1: Comparison: SAFO Worn vs SAFO Not Worn; Paired Wilcoxon Sign Rank TEst; Test type: Superiority or Other; p > .54, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: SAFO Worn vs SAFO Not Worn; Test type: Superiority or Other; p = 0.20, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Groups:
- SAFO Worn: SAFO worn: Child wears their prescirbed SAFO for 14 dyas by random assignment
- SAFO Not Worn: SAFO not worn: Child does ont wear their prescribed SAFO for 14 days by random assignment
Arm/Group | SAFO Worn | SAFO Not Worn
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No